CLINICAL TRIAL: NCT01431859
Title: A Double Blind Placebo Controlled Randomised Trial to Study the Effects of Birch Pollen Specific Immunotherapy (BP-SIT) on the Symptoms of the Oral Allergy Syndrome in Adult Patients
Brief Title: Can we Help People With the Oral Allergy Syndrome Eat Fresh Fruit?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Sussex County Hospital (Other)
Responsible Party: Principal Investigator, Nicola Gray, Clinical Research Fellow, Royal Sussex County Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10/143/FREW; 2011-004078-26 (EudraCT Number)
Record Dates: First submitted 2011-09-05; First posted 2011-09-12 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Oral Allergy Syndrome
Keywords: pollen; allergy; food; immunotherapy
MeSH Terms: conditions — Oral Allergy Syndrome; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous injection of placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Birch pollen immunotherapy (Active Comparator)
  Interventions: Biological: Allergovit Birch pollen

INTERVENTIONS:
Biological: Allergovit Birch pollen — Birch pollen specific immunotherapy. Once weekly injection for 7 weeks prior to birch pollen season for 2 consecutive seasons
  Arms: Birch pollen immunotherapy
Other: Placebo — Placebo injection to be given subcutaneously once weekly for 7 weeks prior to birch pollen season for 2 consecutive years.
  Arms: Subcutaneous injection of placebo

SUMMARY:
Birch pollen allergy is increasingly common. It causes asthma and early season hay fever. This is because the body recognises birch pollen and reacts to it, leading to symptoms. Many patients with birch allergy get an itchy and/or swollen mouth when they eat fresh fruit (apples, pears, peaches, plums etc). Some fruit proteins have a similar structure to birch pollen; because of this the body recognises these proteins too causing the immune system to respond. This response causes symptoms of itch and swelling inside the mouth and throat. the investigators want to find out whether it is possible to get rid of the fruit-induced symptoms by using a desensitisation procedure that has been developed for treating the kind of hay fever that is caused by birch pollen. Desensitisation involves giving a small injection of pollen just under the skin and gradually increasing the amount each week. This allows the body to build up a "tolerance" to the injected protein. When the pollen is then encountered in real life the immune system reacts less vigorously so symptoms are less severe. This treatment does reduce hay fever symptoms. Our study aims to find out if this tolerance is transferred to the fruit proteins enabling patients to eat apples with minimal symptoms. Patients will be given apple to eat in a hidden form before treatment and their response assessed. They will then receive either active or dummy pollen injections before birch pollen season. A few months after completing these injections they will have another disguised apple test to see whether their symptoms are any better. If symptoms have improved with treatment then this therapy could be offered to patients in the future. This would allow them to eat fresh fruit without worrying about unpleasant symptoms and improve their hay fever symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age 18 with no upper age limit
* History of typical fruit-related symptoms on eating apples plus or minus other plant-derived foods known to be involved in the pollen-food syndrome
* History of spring rhinitis hay fever
* Positive skin prick test to birch pollen
* Positive open food challenge to apple

Exclusion Criteria:

* Significant medical conditions that may affect the risks of giving BP-SIT (especially uncontrolled asthma or ongoing need for beta-blockers)
* History of moderate to severe systemic reaction to apple, defined as any of: generalised urticaria, generalised angioedema, history convincing for laryngeal oedema, collapse
* Current immunological disease (auto-immune or thyroid disease, immunodeficiency)
* Malignant disease within the past five years (Patients with previous malignant disease that is considered cured, may be included subject to the consent of their oncologist)
* Inability to attend regularly for injections and follow-up visits
* Severe atopic dermatitis
* Previous immunotherapy with birch pollen extract
* Pregnant or not using adequate contraception (post-menopausal, surgically sterilised, long-term abstinent, or barrier methods plus spermicide)
* Breast-feeding
* Evidence of current drug or alcohol misuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change in threshold for eating uncooked apple from baseline, compared to 1 year and 2 years following the intervention. | baseline, 1 year and 2 years
  Baseline measurements will be taken in Winter 2012 assessing the tolerance to fresh apple in a double blind placebo controlled manner. The intervention will start in January 2013.
  Outcomes will be assessed using the double blind placebo controlled food challenge technique in Winter 2013 and 2014. (1 and 2 years after baseline assessment)

SECONDARY OUTCOMES:
Change in symptoms of rhinoconjunctivitis immediately after the first season of immunotherpay compared to 2 seasons of immunotherapy treatment. | baseline, 1 year and 2 years
  Diary cards will be given to patients to complete in the first season following immunotherapy, to assess hay fever symptoms.
Change in conjunctival provocation tests from baseline. | baseline, 1 year and 2 years
  Conjunctival provocation testing will take place at baseline in Winter 2012 using standard birch pollen exracts. Repeat tests will occur Winter 2013 and 2014 to assess changes following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Frew, MBBS MD FRCP, Principal Investigator — Brighton and Sussex University Hospital Trust
Locations (1):
- Royal Sussex County Hospital, Brighton, East Sussex, United Kingdom